CLINICAL TRIAL: NCT00452504
Title: Ascending Single Dose Study of the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of SRA-444 Administered Orally to Healthy Adult Subjects
Brief Title: Single Ascending Dose Study of SRA-444 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 3197A1-100
Record Dates: First submitted 2007-03-23; First posted 2007-03-27 (Estimated); Last update posted 2007-12-05 (Estimated); Status verified 2007-12

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

INTERVENTIONS:
Drug: SRA-444

SUMMARY:
This is a first-in-humans study of SRA-444. This study will provide an initial assessment of the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of SRA-444 (SR formulation) after administration of ascending single oral doses to healthy adult subjects.

ELIGIBILITY:
Inclusion criteria:

* Healthy men or women of nonchildbearing potential aged 18 to 50 years,
* Body mass index in the range of 18 to 30 kg/m2 and body weight ≥50 kg.

Exclusion criteria:

* Family history of sudden death and/or QT prolongation.
* An automatic ECG corrected QT (QTc) interval reading at screening >450 ms and >470 ms for male and female subjects, respectively.
* Sinus bradycardia at screening, defined as a resting heart rate ≤45 bpm. Resting supine blood pressure at screening <110 mm Hg (systolic) and/or <60 mm Hg (diastolic).

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2007-02; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Assessment of the safety and tolerability of SRA-444

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer; Trial Manager, Principal Investigator — For Netherlands, trials-NL@wyeth.com
Locations (1):
- Zuidlaren, Netherlands